CLINICAL TRIAL: NCT03908216
Title: Evaluation of Non-pharmacological and Pharmacological Treatment for Overweight and Obesity in Patients With Cardiovascular Diseases or With High Cardiovascular Risk According to the Results of Patients' Interviews Within the Outpatient Registry
Brief Title: Evaluation of Non-pharmacological and Pharmacological Treatment for oVerweight and Obesity in pAtients of the Outpatient Register (EVA)
Acronym: EVA
Status: Completed | Type: Observational
Sponsor: National Research Center for Preventive Medicine (Other Government)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Other Study IDs: EVA
Record Dates: First submitted 2019-04-06; First posted 2019-04-09 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Overweight and Obesity
Keywords: overweight,obesity,patients' survey,drug&non-drug treatment
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective non-interventional single-centre study aimed to assess the current practice of non-pharmacological treatment and pharmacological therapy of overweight and obesity in patients with cardiovascular diseases (CVD) or with a high risk of CVD according to the patients' survey data

DETAILED DESCRIPTION:
To interview 300 patients with a body mass index (BMI) ≥25 kg / m² of the outpatient register, who come for a primary or secondary visit to the Center. The specifically designed questionnaire contains topics about patients' self-concept of their body mass; doctors' prescriptions of therapy for obesity, patients' adherence to recommendations.

A repeated short telephone interview of these patients will be conducted in 1-1.5 years after visit inclusion to clarify the dynamics of weight and methods of its correction.

ELIGIBILITY:
Inclusion Criteria:

patients of the outpatient "PROFILE" registry with CVD or with a high risk of CVD (≥5%), with overweight (BMI≥25 kg/m2) or obesity (BMI≥30 kg/m2). Presence of written informed consent to participate in the study, fill in the original questionnaire and given consent to the processing of personal data

Exclusion Criteria:

normal weight, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with overweight or obesity and with CVD or with a high risk of CVD
Sampling Method: Non-Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2021-04-03 (Actual); Study Completion 2021-04-03 (Actual)

PRIMARY OUTCOMES:
The proportion of patients received non-pharmacological treatment recommendations | on enrollment
  Non-pharmacological methods of treatment: diet treatment, increasing physical activity
The proportion of patients received pharmacological treatment recommendations | on enrollment
  Anti-obesity drug treatment prescribing
Patients' self-concept of their body mass | on enrollment
  The proportion of patients who assess their weight as normal weight, overweight or obesity. Patient knowledge of obesity and overweight treatment methods

SECONDARY OUTCOMES:
Effect of overweight and obesity treatment | April, 2019 - November, 2020
  Dynamics of the patient's body weight in a prospective observation
Patient self-assessment of previous overweight and obesity treatments effectiveness | April, 2019 - November, 2020
  The proportion of patients who rated the effectiveness of treatment as effective short-term, effective long-term, ineffective

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Yu Martsevich, MD, PhD, Principal Investigator — National Research Center for Preventive Medicine, Moscow, Russia, 101990
Locations (1):
- Yulia Lukina, Moscow, Russia